CLINICAL TRIAL: NCT03856736
Title: Effects of Aerobic Exercise on Telomere Length in Patients With Systolic Heart Failure: A Randomized Clinical Trial.
Brief Title: Aerobic Exercise and Telomere Length in Patients With Heart Failure.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 180651
Record Dates: First submitted 2019-02-15; First posted 2019-02-27 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Telomere Length; Aerobic Exercise
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIAT (Experimental): Composite of the execution of moderated-intensity aerobic training (MIAT) twice week.
  Interventions: Other: MIAT; Other: Control
- Control (Experimental): Consisting of two session per week of different activities, such as body relaxation, low-intesity/volume of aerobic exercise to mimic sham group.
  Interventions: Other: MIAT; Other: Control

INTERVENTIONS:
Other: MIAT — Moderated aerobic exercise
Other: Control — Weekly body relaxation and sham group

SUMMARY:
The present study will analyze and compare the chronic effects of aerobic exercise in subjects with systolic heart failure on telomere length.

DETAILED DESCRIPTION:
Aging can be characterized by an organic and functional decrease, which is not related to disease, that is, a process that happens naturally over time. One of the markers of the aging process is telomeres, which consist of a complex of DNA sequences located at the ends of the chromosome, composed of protective proteins that have the function of protecting information from the DNA (genome), that is, telomeres are responsible for reconstructing the information lost during cell division due to the wear and tear of the chromosome ends. The telomere length may be shorter in some diseases, such as heart failure with reduced ejection fraction (HFREF) compared with healthy subjects.

The HFREF is a complex clinical syndrome of poor prognosis and high prevalence. Its characteristics include fatigue, dyspnea and intolerance to physical exertion due to reduction in cardiac output, concomitant with respiratory changes, weakness in peripheral muscles and incidence of depression. Exercise as a strategy for the treatment of heart failure (HF) can be effective in improving the quality of life, functional capacity and prognosis of the disease. In sedentary individuals who do not have HF, a natural reduction of telomeres occurs, which is associated with the early development of the aging process. Increasing or maintaining the size of telomeres can be a way to intervene in the aging process and thus slow the progression of HF, since one of its main functions is to protect the chromosome from cellular aging.

One of the most promising strategies for intervening in aging is the practice of physical exercise. However, the effects of physical exercise on the telomere length of individuals with HF are unknown. However, we know that physical exercise for HF shows positive results in relation to functional capacity, as measured by peak oxygen consumption (VO2peak). In addition, the improvement in functional capacity, increase in peak oxygen consumption (VO2peak), is directly related to the increase in telomere length. However, there is a lack of concise results in the literature regarding the chronic effects of aerobic exercise on the telomere length in subjects with HFREF.

Therefore, the aim of the present study will be to analyze and compare the chronic effects of aerobic exercise in subjects with HFREF on telomere length.

The specifics aims of this study are: to analyze and compare the chronic effects of aerobic exercise in individuals with HFREF in the following variables: Functional Capacity (Cardiopulmonary Exercise Testing); Echocardiographic Variables by Doppler echocardiogram; Endothelial Function measured by Flow-Mediated Dilation (FMD) of the Brachial Artery; Walking Ability measured by a Self-Selected Walking Speed Test (SSWST)

This is a randomized clinical trial, with two intervention groups that will be assessed pre and post intervention. The randomization sequence will be generated by REDCap and it will be performed by a participant not involved in the other study phases (principal investigators will be blinded).

For significance level of 5%, power of 80%, difference to be detected equal to the standard deviation of 0.0026, the sample size calculated is 10 patients for each group (20 in total). Considering 20% loss, it will be necessary to include 12 patients per group (24 patients in total).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of HF with ejection fraction <40%;
* Clinically stable patients with at least three months on optimal HF treatment;
* Age between 50 and 80 years;
* New York Heart Association (NYHA) functional class II to III;
* No contraindications to participate in an exercise program;
* Mentally able to understand instructions during the study.

Exclusion Criteria:

* Severe valve disease;
* Peripheral artery disease with symptoms of intermittent claudication;
* Uncontrolled hypertension;
* Drug or alcohol abuse;
* Cognitive and/or osteomyoarticular conditions that prevent exercise;
* Logistical impossibility of attending the hospital intervention;
* Engaging in supervised physical exercise in the past three months;
* Do not complete the run-in period.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Biological Aging | 16 weeks
  Telomere Length

SECONDARY OUTCOMES:
Aerobic Capacity | 16 weeks
  Cardiopulmonary Exercise Test - VO2peak
Echocardiography Variables | 16 weeks
  Differents echocardiography variables such as Strain Global Longitudinal
Endothelial Function | 16 weeks
  Flow-mediated dilation (FMD) of Brachial Artery
SSWS | 16 weeks
  Walking Ability measured by a Self-Selected Walking Speed Test (SSWST)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Stein, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Franzoni LT, Garcia EL, Motta SB, Ahner MM, Bertoletti OA, Saffi MAL, da Silveira AD, Pereira AA, Pereira AH, Danzmann LC, Stein R. Aerobic exercise and telomere length in patients with systolic heart failure: protocol study for a randomized controlled trial. Trials. 2022 Apr 11;23(1):283. doi: 10.1186/s13063-022-06257-1. PMID 35410445